CLINICAL TRIAL: NCT04057456
Title: Cannabinoids and an Anti-inflammatory Diet for the Treatment of Neuropathic Pain After Spinal Cord Injury
Acronym: CATNP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eldon Loh, MD (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Responsible Party: Sponsor-Investigator, Eldon Loh, MD, Physician, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 6465
Record Dates: First submitted 2019-08-01; First posted 2019-08-15 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
Keywords: Nabilone; Spinal Cord Injury; Neuropathic pain; Pain; Anti Inflammatory Diet
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia; Pain | interventions — nabilone

STUDY DESIGN:
Intervention Model Description: Eligible participants who consent to study participation will be randomized to one of four groups: 1) Nabilone and Placebo Diet, 2) Placebo Capsule and Anti-inflammatory Diet, 3) Nabilone and Anti-inflammatory Diet, and 4) Placebo Capsule and Placebo Diet. Following randomization, participants will begin a study agent titration period (nabilone or placebo) in order to determine a safe and effective nabilone dose for each participant. Once the appropriate nabilone (or placebo) dosage for each participant is determined, participants will begin their respective interventions over the course of the 4-week treatment period. All outcome measures will be at assessed baseline, after the study agent titration period, and post-testing (following the 4-week treatment period).
Who Masked: Participant, Care Provider, Investigator
Masking Description: No other parties will be masked for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo diet and placebo capsules (Placebo Comparator): Participants taking the placebo diet and capsules
  Interventions: Other: Placebo diet; Other: Placebo capsules
- Placebo diet and Nabilone capsules (Active Comparator): Capsules will be 0.5mg nabilone. Participants will take up to 8 capsules per day for a maximum dose of 4mg of nabilone per day.
  Interventions: Other: Placebo diet; Drug: Nabilone Capsules
- Anti-inflammatory diet and placebo capsules (Active Comparator): This meal plan will eliminate foods that have been established as pro-inflammatory (e.g. processed foods, refined sugars, refined wheat products, etc.) as well as foods that are commonly associated with even mild intolerances (e.g. cow's milk) and those that negatively impact cardiovascular health (e.g. hydrogenated oils, alcohol, coffee, refined sugars and wheat, trans fats, processed foods). In their place, the meal plan will consist of foods with established anti-inflammatory properties (e.g. (Oily fish, lean poultry, dark leafy greens, cruciferous vegetables, nuts, whole grains, most kinds of berries, etc).
  Interventions: Other: Anti-inflammatory diet; Other: Placebo capsules
- Anti-inflammatory diet and Nabilone capsules (Active Comparator): Capsules will be 0.5mg nabilone. Participants will take up to 8 capsules per day for a maximum dose of 4mg of nabilone per day.
  This meal plan will eliminate foods that have been established as pro-inflammatory (e.g. processed foods, refined sugars, refined wheat products, etc.) as well as foods that are commonly associated with even mild intolerances (e.g. cow's milk) and those that negatively impact cardiovascular health (e.g. hydrogenated oils, alcohol, coffee, refined sugars and wheat, trans fats, processed foods). In their place, the meal plan will consist of foods with established anti-inflammatory properties (e.g. (Oily fish, lean poultry, dark leafy greens, cruciferous vegetables, nuts, whole grains, most kinds of berries, etc).
  Interventions: Other: Anti-inflammatory diet; Drug: Nabilone Capsules

INTERVENTIONS:
Other: Placebo diet — The dietitian will assist in developing a diet that is isocaloric to the anti-inflammatory diet and healthy (for the sake of the participants' well-being, and to blind participants), while allowing many foods that are (counterintuitively) pro-inflammatory (e.g. whole wheat bread, white beans, oats, soy, eggplant, raspberries, pumpkin seeds, popcorn, etc). Occasional "cheat" foods are built into the placebo diet but with more pro-inflammatory options (e.g. two glasses of wine per week).
  Arms: Placebo diet and Nabilone capsules; Placebo diet and placebo capsules
Other: Anti-inflammatory diet — Participants will also be given a list of foods that they are allowed on the anti-inflammatory diet, and a list of foods to avoid so that they can make informed substitutions to the meals and ingredients that they are given. The study participants will be given a one-week meal plan with accompanying recipes. Occasional "cheat" foods are built into the anti-inflammatory diet (e.g. two bottles of beer per week)
  Arms: Anti-inflammatory diet and Nabilone capsules; Anti-inflammatory diet and placebo capsules
Drug: Nabilone Capsules — Capsules will be 0.5mg nabilone. Participants will undergo a 5-week titration period by taking 1 (0.5mg) nabilone capsule per day for a three-day period. The dose will be increased on a fixed schedule by 1 (0.5mg) capsule every three days to a maximum of 8 capsules/day (4mg). Dosage will be maintained if higher doses are not tolerated or if sufficient relief is obtained (at least a 2-point change on the NRS). Once the appropriate nabilone (or placebo) dosage for each participant is determined, participants will begin their respective interventions over the course of the 4-week treatment period.
  Arms: Anti-inflammatory diet and Nabilone capsules; Placebo diet and Nabilone capsules
Other: Placebo capsules — Placebo capsules contain no active ingredient. Participants on placebo capsules will undergo the same 5-week titration period and intervention period as those on active treatment.
  Arms: Anti-inflammatory diet and placebo capsules; Placebo diet and placebo capsules

SUMMARY:
Neuropathic pain is a common complication following spinal cord injury (SCI) that significantly decreases quality of life. Treatment options are limited, and current treatments can have significant side effects. Those with SCI have identified a need for additional treatment options, particularly those that are not medications. Nabilone and an anti-inflammatory diet are two treatments that may provide pain relief while being better tolerated. This study will evaluate the benefits of these treatments for neuropathic pain after SCI. Study participants will receive either an anti-inflammatory diet or a placebo diet, and nabilone or a placebo for 4 weeks. It is expected that an anti-inflammatory diet and nabilone will significantly decrease pain intensity and improve function. The combination of both treatments together is expected to have a greater effect than each alone.

DETAILED DESCRIPTION:
Nabilone and an anti-inflammatory diet are two novel treatments that may be beneficial for managing Neuropathic Pain (NP) after Spinal Cord Injury (SCI).

Neuropathic pain is a common complication following SCI that significantly decreases quality of life. Treatment options are limited, and current treatments can have significant side effects. Those with SCI have identified a need for additional treatment options, particularly those that are not medications. Cannabinoids and an anti-inflammatory diet may provide pain relief while being better tolerated.

The Co- Sponsor Investigators will test the potential benefits of these treatments for neuropathic pain after SCI.

Clinically, cannabinoids have been shown to be effective in the management of central NP after multiple sclerosis (MS), and although they have been trialed for a variety of complications after SCI, direct evidence for their ability to manage NP in this population is limited. Further, no studies have evaluated the efficacy of synthetic cannabinoids (nabilone) for the treatment of NP after SCI. Accordingly, the CanPainSCI Clinical Practice Guidelines concluded that the evidence is insufficient to develop a specific recommendation regarding cannabinoids in the treatment of NP after SCI. In addition, relevant side effects for those with SCI have not been well documented. Despite this, cannabinoids have been increasingly used as a treatment option for NP after SCI, particularly given increased access to, and greater societal acceptance of, cannabinoids in general. Studies that evaluate the effectiveness and side effects of cannabinoids and synthetic cannabinoids in the SCI population are therefore urgently needed.

An anti-inflammatory diet has recently shown promise in the management of NP after SCI. An RCT comparing an anti-inflammatory diet to placebo identified a reduction in sensory NP symptoms following SCI. This RCT was done in a general population of SCI patients and did not necessarily select those who were experiencing significant neuropathic pain. Therefore, additional evidence to demonstrate treatment effect will be important to justify widespread adoption of this diet for NP after SCI.

The study will collect data on a sample of up to 140 patients with SCI and at- and/or below-level neuropathic pain >3/10 in severity on the numeric rating scale.

The Principal Investigators will assess the treatment's effects on quality of life and pain management. If the study is successful, the results (and an evaluation of the process) will be used to inform an affordable and sustainable anti-inflammatory nutrition program to be implemented at Power Cord. This nutrition program will also be widely disseminated and potentially act as a template for similar programs In SCI care centres across Canada.

This study will assess blood samples at three time points for analysis of pro and anti-inflammatory markers. The research coordinator (blinded to the randomization) will assess patients using various quality of life and pain assessment questionnaires during clinic visits, at home or by telephone interview.

The type, level, and completeness of injury will be documented, and, if necessary, updated at each in-person visit. Each participant will be provided with instructions and study schedule. Protocol compliance will be tested through product count and interviews at each follow-up visit. Side effects will be assessed using standardized case report forms at each visit. Study visits may be in person or over the phone. Participants will be encouraged to report any events they may experience directly to the coordinator.

Participants who withdraw consent to continue treatments, will be encouraged to undergo the planned assessments. Withdrawal at the request of investigators or medical personnel may include, but are not limited to:

1. Symptoms are deemed to be potentially related to the study product
2. New diagnosis of exclusion criteria;
3. Unacceptable side effects;
4. Death

Estimated time to complete recruitment: Averaging 36 months, approximately 3 years.

ELIGIBILITY:
Inclusion:

1. Age 25 and over, based on year of birth
2. Signed informed consent obtained prior to any study-related activities
3. BMI 18-40
4. A spinal cord injury at least 12 months duration, nonprogressive for at least 6 months
5. At- and/or below-level neuropathic pain >3/10 in severity on the numeric rating scale (NRS) (below-level neuropathic pain will be defined as pain >1 dermatomal level below the neurologic level of injury). Participants will need an average >3/10 pain over the past 7 days on screening, and to complete a daily diary for the week prior to randomization in the morning with an average pain severity of >3/10 on at least 4 diary entries.
6. Ongoing constant pain for at least 3 months, or relapsing/remitting pain for at least 6 months.
7. Dosing of other pain medications (NSAIDs, opioids, non-opioid analgesics, anti-epileptic drugs, antidepressants) should be stable for at least 1 month prior to study entry.
8. Any cannabinoids, or cannabinoid medications (e.g. nabilone) will need to be stopped at least 1 month prior to screening for and inclusion in the study.
9. Females of childbearing potential must agree to use a medically approved method of birth control (e.g. hormonal contraceptives, intrauterine devices, vasectomy/tubal ligation, barrier methods and double-barrier method) and must have a negative pregnancy test results at screening and baseline.

Exclusion:

1. History of psychotic disorder
2. History of convulsive disorders
3. History of substance abuse
4. experienced myocardial infarction or clinically significant cardiac dysfunction within the last 12 months
5. Significantly impaired hepatic function at Visit A1 or B1 (Alanine aminotransferase [ALT] >5 upper limit of normal [ULN] or total bilirubin [TBL] >2 ULN) OR the ALT or Aspartate aminotransferase (AST) >3 ULN and TBL >2 ULN (or international normalized ratio [INR] >1.5)
6. Female patients of child bearing potential and male patients whose partner is of child bearing potential, unless willing to ensure that they or their partner use effective contraception, during the study and for three months thereafter
7. Female patient who is pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter
8. Current suicidal ideation
9. Current use of cannabinoids or cannabinoid medication
10. Intolerance to cannabinoids
11. Traumatic SCI superimposed on prior congenital stenosis
12. Preexisting myelopathy of other causes (e.g. transverse myelitis, epidural abscess, congenital spondylotic myelopathy)
13. Presence of other neurologic conditions, medical conditions or pain that could confound the assessment of neuropathic pain after SCI
14. Currently enrolled in another clinical trial
15. Any other significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, may influence the result of the study, or affect the patient's ability to participate in the study
16. Following a physical examination, the patient has any abnormalities that, in the opinion of the investigator would prevent the patient from safe participation in the study

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Average pain intensity | Baseline and 9 weeks
  Change from baseline to end of study in average pain intensity evaluated using the Numeric Rating Scale, which measures pain using a scale of 1-10 (1 being mild, and 10 being severe)
Sensory changes | Baseline and 9 weeks
  Changes from baseline to end of study in the items on the Neuropathic Pain Questionnaire
Pain relief | Baseline and 9 weeks
  Proportion of participants achieving at least 30% and 50% pain relief between treatments.

SECONDARY OUTCOMES:
Patient global impression of change | Baseline and 9 weeks
  Change from first study visit to end of study in the patient global impression of change questionnaire
Financial feasibility of following anti-inflammatory diet | 9 weeks
  This will be analyzed using a cost estimate created by the study team, and will be compared to the Productivity Costs Questionnaire which assesses participant's income.
Mood Centre for Epidemiologic Studies-Depression scale | Baseline and 9 weeks
  Changes from baseline to end of study in mood, assessed by the Mood Centre for Epidemiologic Studies Depression Scale, which has 20 questions that can be answered using four options: Rarely, Some or a little of the time, Occasionally, and Most or all of the time.
Sleep | Baseline and 9 weeks
  Changes from baseline to end of study in sleep assessed by Leeds Sleep Evaluation Questionnaire
Spasticity | Baseline and 9 weeks
  Changes from baseline to end of study in spasticity documented using the SCI-Spasticity Evaluation Tool (SCI-SET)
Pro-Inflammatory biomarkers | Baseline and 9 weeks
  Changes from baseline to end of study in blood inflammatory biomarkers interleukin-2 (IL-2), IL-6, IL-1β, tumor necrosis factor alpha (TNF-α), interferon gamma (IFN-γ) and prostaglandin E2 (PGE2) will be evaluated through blood collection and analysis using an ELISA analysis.
Profile of Mood States | Baseline and 9 weeks
  Change from baseline to end of study in Profile of Mood States questionnaire, this questionnaire evaluates what different types of moods the participant has felt and rates each mood into 5 possible answers: Not At All, A Little, Moderately, Quite a lot, Extremely.
Anti-Inflammatory Biomarkers | Baseline and 9 weeks
  Changes from baseline to end of study in blood anti-inflammatory biomarkers IL-4, IL-10 and IL-1a will be evaluated through blood collection and analysis using an ELISA analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Eldon Loh, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; David Ditor, MD, Principal Investigator — Brock University
Locations (1):
- St. Joseph's Health Care London - Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loh E, Guy SD, Mehta S, Moulin DE, Bryce TN, Middleton JW, Siddall PJ, Hitzig SL, Widerstrom-Noga E, Finnerup NB, Kras-Dupuis A, Casalino A, Craven BC, Lau B, Cote I, Harvey D, O'Connell C, Orenczuk S, Parrent AG, Potter P, Short C, Teasell R, Townson A, Truchon C, Bradbury CL, Wolfe D. The CanPain SCI Clinical Practice Guidelines for Rehabilitation Management of Neuropathic Pain after Spinal Cord: introduction, methodology and recommendation overview. Spinal Cord. 2016 Aug;54 Suppl 1:S1-6. doi: 10.1038/sc.2016.88. PMID 27444714
- [Background] Guy SD, Mehta S, Casalino A, Cote I, Kras-Dupuis A, Moulin DE, Parrent AG, Potter P, Short C, Teasell R, Bradbury CL, Bryce TN, Craven BC, Finnerup NB, Harvey D, Hitzig SL, Lau B, Middleton JW, O'Connell C, Orenczuk S, Siddall PJ, Townson A, Truchon C, Widerstrom-Noga E, Wolfe D, Loh E. The CanPain SCI Clinical Practice Guidelines for Rehabilitation Management of Neuropathic Pain after Spinal Cord: Recommendations for treatment. Spinal Cord. 2016 Aug;54 Suppl 1:S14-23. doi: 10.1038/sc.2016.90. PMID 27444715
- [Background] Allison DJ, Thomas A, Beaudry K, Ditor DS. Targeting inflammation as a treatment modality for neuropathic pain in spinal cord injury: a randomized clinical trial. J Neuroinflammation. 2016 Jun 17;13(1):152. doi: 10.1186/s12974-016-0625-4. PMID 27316678
- [Background] Fine PG, Rosenfeld MJ. Cannabinoids for neuropathic pain. Curr Pain Headache Rep. 2014 Oct;18(10):451. doi: 10.1007/s11916-014-0451-2. PMID 25160710
- [Background] Nielsen S, Germanos R, Weier M, Pollard J, Degenhardt L, Hall W, Buckley N, Farrell M. The Use of Cannabis and Cannabinoids in Treating Symptoms of Multiple Sclerosis: a Systematic Review of Reviews. Curr Neurol Neurosci Rep. 2018 Feb 13;18(2):8. doi: 10.1007/s11910-018-0814-x. PMID 29442178
- [Background] Eisenstein M. Medical marijuana: Showdown at the cannabis corral. Nature. 2015 Sep 24;525(7570):S15-7. doi: 10.1038/525S15a. No abstract available. PMID 26398734
- [Background] Langford RM, Mares J, Novotna A, Vachova M, Novakova I, Notcutt W, Ratcliffe S. A double-blind, randomized, placebo-controlled, parallel-group study of THC/CBD oromucosal spray in combination with the existing treatment regimen, in the relief of central neuropathic pain in patients with multiple sclerosis. J Neurol. 2013 Apr;260(4):984-97. doi: 10.1007/s00415-012-6739-4. Epub 2012 Nov 21. PMID 23180178
- [Background] Mucke M, Phillips T, Radbruch L, Petzke F, Hauser W. Cannabis-based medicines for chronic neuropathic pain in adults. Cochrane Database Syst Rev. 2018 Mar 7;3(3):CD012182. doi: 10.1002/14651858.CD012182.pub2. PMID 29513392
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Ware MA. Medical Cannabis Research: Issues and Priorities. Neuropsychopharmacology. 2018 Jan;43(1):214-215. doi: 10.1038/npp.2017.222. No abstract available. PMID 29192670
- [Background] Karschner EL, Darwin WD, McMahon RP, Liu F, Wright S, Goodwin RS, Huestis MA. Subjective and physiological effects after controlled Sativex and oral THC administration. Clin Pharmacol Ther. 2011 Mar;89(3):400-7. doi: 10.1038/clpt.2010.318. Epub 2011 Feb 2. PMID 21289620
- [Background] De Gregorio D, McLaughlin RJ, Posa L, Ochoa-Sanchez R, Enns J, Lopez-Canul M, Aboud M, Maione S, Comai S, Gobbi G. Cannabidiol modulates serotonergic transmission and reverses both allodynia and anxiety-like behavior in a model of neuropathic pain. Pain. 2019 Jan;160(1):136-150. doi: 10.1097/j.pain.0000000000001386. PMID 30157131
- [Background] Margolis JM, Juneau P, Sadosky A, Cappelleri JC, Bryce TN, Nieshoff EC. Health care resource utilization and medical costs of spinal cord injury with neuropathic pain in a commercially insured population in the United States. Arch Phys Med Rehabil. 2014 Dec;95(12):2279-87. doi: 10.1016/j.apmr.2014.07.416. Epub 2014 Aug 24. PMID 25159715
- [Background] Serpell M, Ratcliffe S, Hovorka J, Schofield M, Taylor L, Lauder H, Ehler E. A double-blind, randomized, placebo-controlled, parallel group study of THC/CBD spray in peripheral neuropathic pain treatment. Eur J Pain. 2014 Aug;18(7):999-1012. doi: 10.1002/j.1532-2149.2013.00445.x. Epub 2014 Jan 13. PMID 24420962
- [Background] Siddall PJ, Cousins MJ, Otte A, Griesing T, Chambers R, Murphy TK. Pregabalin in central neuropathic pain associated with spinal cord injury: a placebo-controlled trial. Neurology. 2006 Nov 28;67(10):1792-800. doi: 10.1212/01.wnl.0000244422.45278.ff. PMID 17130411